CLINICAL TRIAL: NCT02305290
Title: Outcomes of Endoscopic Resection in the Upper Gastrointestinal Tract
Brief Title: Upper GI Outcomes Following EMR
Acronym: UGI-EMR
Status: Completed | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: HREC2014/7/4.6 (4033)
Record Dates: First submitted 2014-07-30; First posted 2014-12-02 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Adenoma, Villous
MeSH Terms: conditions — Adenoma, Villous | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopic Mucosal Resection: Patients who are referred for Endoscopic Mucosal Resection of Upper Gastrointestinal Lesions will be included in this cohort.
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection

SUMMARY:
The purpose of this study is to evaluate the long-term outcomes of Endoscopic Resection (ER) of superficial lesions of the Upper Gastrointestinal Tract(UGIT)

DETAILED DESCRIPTION:
Endoscopic resection (ER) of superficial lesions of the upper gastrointestinal tract is a safe and effective surgery-sparing modality in experienced hands. It is often curative of dysplastic lesions and is associated with minimal complications and high patient acceptance (1-5). Westmead Hospital has accumulated a significant amount of experience in the removal of such lesions; however, there is limited research to document the long term outcomes of patients undergoing endoscopic resection.The purpose of this study is to evaluate the long-term outcomes of ER of superficial lesions of the UGIT.

ELIGIBILITY:
Inclusion Criteria:

* UGIT lesion > 10mm
* Lesion limited to the mucosal and/or submucosal layer (T1 lesion)
* Aged 18 years or older

Exclusion Criteria:

* Lesion less than 10mm
* Gastric lesion involves the muscularis propria (T2 lesion) on other staging modalities such as endoscopic ultrasonography (EUS)
* Aged younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have Upper Gastrointestinal Tract adenomas which are amendable to Endoscopic Mucosal Resection
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Observed procedural data | 14 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability Outcomes

SECONDARY OUTCOMES:
Analysis of the costs of this procedure compared to previous treatments | 14 days
  Perform cost-utility analyses comparing different treatment approaches for UGIT lesions

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia